CLINICAL TRIAL: NCT05503628
Title: The Validity and Reliability of the Trunk Impairment Scale-modNV and the AMTI AccuGait Optimized Force Platform Across Mild and Moderate Disability Levels in the MS Population
Brief Title: A Measurement Study of TIS-modNV and AccuGait Force Platform in People With MS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nordlandssykehuset HF (Other)
Collaborators: Nord University (Other); Helse Nord (Industry)
Responsible Party: Sponsor
Other Study IDs: Trunk & balance tests in MS; HNF1608-21 (Other Grant/Funding Number: Northern Norway Regional Health Authoroty)
Record Dates: First submitted 2022-08-15; First posted 2022-08-16 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Trunk control; Balance; Outcome measure
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The current project will fill a knowledge gap in the follow-up of people with Multiple Sclerosis (MS) with mild and moderate disability levels, with the purpose to assess the adequacy of measurement tools for trunk control and balance, functions that are pre-requisites for optimal performance in everyday physical activities.

DETAILED DESCRIPTION:
Trunk control and balance, necessary for daily activities, are frequently impaired in people with MS. Adequate measurement tools for clinical- and research purposes are thus warranted. In this study two measurement tools will be explored:

1. The Trunk Impairment scale - modified Norwegian version (TIS-modNV), which has demonstrated high validity and reliability in individuals with stoke (Gjelsvik et al., 2012), however its properties has not yet been assessed in people with MS. Concurrent validity with a balance scale, the Mini-Balance Evaluation Systems Test (Mini-BESTest), will be assessed as well as its inter- and intra-rater reliability.
2. The AMTI Accugait Optimized™ multi-axis force platform (AMTI, Inc., Newton, MA) will be examined as there is a lack of studies measuring its properties within the MS population. A validity assessment of this tool will be included in this measurement study.

This study is two-parted, each with a separate aim:

Aim part 1: To determine the validity and reliability of the TIS-modNV across mild and moderate disability levels in the MS population.

Aim part 2: To determine the concurrent validity of the AMTI AccuGait OptimizedTM force plate system compared to the Mini-BESTest across mild and moderate disability levels in the MS population.

ELIGIBILITY:
Inclusion Criteria:

* MS diagnosis (McDonalds criteria)
* EDSS= 0-6.5
* Ability to walk minimum 6 meters

Exclusion Criteria:

* People will be excluded if not being able to follow test instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted in Bodø, Nordland county, Norway involving the MS population affiliated to the MS-outpatient clinic at Nordland Hospital (NLSH) and whose adress is in one of the eight municipalities in the Salten region. All people in this population, fitting the inclusion criteria will be requested to participate. People covering the whole range of EDSS 0-6.5 will be recruited. If too many people consents to participate there will be draw.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-08-15 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
The modified Trunk Impairment Scale - Norwegian version (TIS-modNV) | 01 January 2023
  TIS-modNV is a six-item ordinal scale measuring impairments of trunk control. The total score ranges between 0-16, where 16 is the best score in trunk control. The scale is developed for and valid and reliable for people with stroke.
AMTI AccuGait OptimizedTM (Advanced Mechanical technology, Inc., Watertown, USA) multi-axis force plate system | 01 January 2023
  Force- platform assessing different domains of balance (ie. centre of pressure, sway) in bi- and unipedal standing with eyes open and with eyes closed.

OTHER OUTCOMES:
The Mini Balance Evaluation Systems Test (Mini-BESTest) | 01 January 2023
  Mini-BESTest is a 14-item ordinal scale, measuring balance in standing and walking. The total scores ranges from 0-28, were 28 is the best score of balance performance. The Norwegian translation of the test is valid and reliable for people with MS.
Expanded Disability Status Scale (EDSS) | 01 January 2023
  EDSS is a method of quantifying and monitoring disability in people with MS on a scale from 0-10 and is widely used in clinic and research. A total score of 0 describes "no disability" and a score 10 describes "death due to MS". EDSS scores 0-6.5 (the levels included in this study) encompasses individuals with normal neurological exam/fully ambulatory (score 0) to individuals requiring a walking aids (cane, crutch) to walk about 20m without resting (score 6.5).

CONTACTS AND LOCATIONS:
Overall Officials: Petter Øyen, PHD, Study Director — Nordlandssykehuset HF
Locations (1):
- Nordland Hospital Trust, Bodø, Norway

IPD SHARING:
Plan to Share IPD: No